CLINICAL TRIAL: NCT04440007
Title: A Phase 2, Open Label, Randomized Study of the Efficacy and Safety of STI-5656 (Abivertinib Maleate) With Standard of Care Versus Standard of Care in Subjects Hospitalized With COVID-19
Brief Title: Study of the Efficacy and Safety of STI-5656 (Abivertinib Maleate) in Subjects Hospitalized With COVID-19
Acronym: SOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STI-5656-2001
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — abivertinib; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abivertinib with Standard of Care (Experimental): STI-5656 (abivertinib maleate) capsule administered orally 200 mg QD up to 28 days or until hospital discharge, in addition to standard of care
  Interventions: Drug: Abivertinib; Other: Standard of Care
- Standard of Care (Active Comparator): Standard of care treatments for COVID-19 as determined appropriate by the Investigator
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Abivertinib — Abivertinib maleate is a third-generation EGFR tyrosine kinase inhibitor and BTK Inhibitor. The starting dose is 200 mg p.o. QD for up to 28 days.
  Other Names: abivertinib maleate; avitinib; AC0010; STI-5656
  Arms: Abivertinib with Standard of Care
Other: Standard of Care — Standard of Care as determined by the Investigator

SUMMARY:
Study to assess the safety and efficacy of STI-5656 (Abivertinib Maleate) plus SOC versus SOC in subjects hospitalized with COVID-19

DETAILED DESCRIPTION:
This is a Phase 2, open-label, randomized 2-arm multicenter study to assess the safety and efficacy of STI-5656 (Abivertinib Maleate) administered orally plus Standard of Care (SOC) versus SOC in hospitalized subjects with RT-PCR confirmed SARS-CoV-2 infection and COVID-19 pneumonia (documented radiographically). Only hospitalized patients are eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed infection with SARS-CoV-2 per World Health Organization (WHO) criteria (including positive RT-PCR nucleic acid test of any specimen [eg, respiratory, blood, urine, stool, or other bodily fluid]) within 7 days of randomization
* Hospitalized with COVID-19 pneumonia (documented radiographically) and oxygen saturation <94% on room air or subject requires supplemental oxygen
* Able to swallow capsules
* Willing to follow contraception guidelines
* Subject or family member/caregiver must have provided written informed consent which includes signing the institutional review board approved consent form prior to participating in any study related activity. However, if obtaining written informed consent is not possible, other procedures as provided in the March 27th, 2020 FDA Guidance on Conduct of Clinical Trials of Medical Products during COVID-19 Pandemic, Question 10, may be used

Exclusion Criteria:

* Known cardio-pulmonary resuscitation within 14 days prior to randomization
* Pregnant or breast feeding
* Suspected uncontrolled active bacterial, fungal, viral, or other infection (besides infection with SARS-CoV-2)
* Alanine aminotransferase (ALT) ≥ 3x upper limit of normal (ULN) and total bilirubin > 2x ULN
* QTcF prolongation >480 milliseconds
* Uncontrolled or untreated symptomatic arrhythmias, myocardial infarction within the last 6 weeks, or congestive heart failure (NYHA Grade 3 or 4). Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening are allowed to enroll
* Treatment with a strong cytochrome P450 (CYP3A4 inhibitor (within 14 days before first dose of study drug) or inducer (within 7 days before first dose of study drug)
* Received anti-rejection or immunomodulatory drugs (eg, anti-cytokines, BTK inhibitors, JAK inhibitors, PI3K inhibitors) within 30 days before randomization on study
* Concurrent participation in another clinical trial involving therapeutic interventions (observational study participation is acceptable)
* Any condition that confounds the ability to interpret data from the study
* Relevant renal impairment (eGFR <60 mL/min)
* Any significant medical condition, laboratory abnormality or psychiatric illness that would interfere or prevent the subject from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD JD, Study Director — Sorrento Therapeutics, Inc.
Locations (6):
- United States (6):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Teradan Clinical Trials, Brandon, Florida
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Clinical Trials of SWLA, Lake Charles, Louisiana
  - Quality Clinical Research, Omaha, Nebraska
  - Memorial Hermann Memorial City Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo With Standard of Care: Oral placebo capsule administered orally QD up to 28 days or until hospital discharge, in addition to standard of care of care treatment for COVID-19 as determined appropriate by the Investigator
  Standard of Care: Standard of Care as determined by the Investigator
Period: Overall Study
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
Started | 48 | 48
Completed | 36 | 36
Not Completed | 12 | 12
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 7 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Inability to draw blood for labs and being transferred to a nursing facility with no transportation | 1 | 2
Not completed — Discontinued prior to dosing | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 59.9 (12.38) | 57.4 (12.88) | 58.6 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 31 | 31 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 37 | 36 | 73
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 11 | 15
  White | 42 | 33 | 75
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 96
Weight [Mean (Standard Deviation); unit: kg] | 101.94 (30.694) | 100.12 (25.855) | 101.03 (28.243)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Alive and Free of Respiratory Failure at Day 28
Description: Percentage of subjects alive and free of respiratory failure at Day 28, where respiratory failure, is defined based on resource utilization of any of the following modalities:
  * Noninvasive positive pressure ventilation or continuous positive airway pressure
  * Endotracheal intubation and mechanical ventilation
  * Oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20L/min with fraction of delivered oxygen ≥ 0.5)
  * Extracorporeal membrane oxygenation
Time Frame: Randomization to Day 28
Population: A total of 48 subjects in the STI-5656 group and 48 subjects in the placebo group were included in the analysis of the primary endpoint in the FAS. For a number of the excluded subjects, the reason for exclusion from the primary endpoint analysis was that they had no baseline value available.
Measure: Count of Participants; unit: Participants
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
Number analyzed (Participants) | 48 | 48
Participants | 40 | 38

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Number of Participants with Treatment-emergent Adverse Events
Time Frame: Randomization through study completion to 94 days
Population: A total of 48 subjects in the STI-5656 group and 46 subjects in the placebo group were included in the analysis of the secondary endpoint in the FAS. For a number of the excluded subjects, the reason for exclusion from the secondary endpoint analysis was that they had no baseline value available. 46 subjects were analyzed for the placebo group as 2 subjects were randomized to the placebo group who ET prior to dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
Number analyzed (Participants) | 48 | 46
Participants | 31 | 23

3. Secondary Outcome: Percentage of Subjects Alive and Free of Respiratory Failure at Day 60
Description: Percentage of subjects alive and free of respiratory failure at Day 60
Time Frame: Randomization to Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
Number analyzed (Participants) | 48 | 48
Participants | 37 | 35

4. Secondary Outcome: Change in C-Reactive Protein (CRP)
Description: Mean change in CRP on Day 7
Time Frame: Day 7
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
Number analyzed (Participants) | 48 | 48
ng/ml | 71.43 (527.102) | 66.67 (755.613)

5. Secondary Outcome: Partial Pressure of Oxygen in Arterial Blood and Fraction of Inspired Oxygen (PaO2/FiO2)
Description: PaO2/FiO2 at Day 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
Number analyzed (Participants) | 48 | 48
mmHG | 210.61 (112.686) | 253.34 (103.679)

6. Secondary Outcome: All-cause Mortality at Day 60 and Day 90
Description: All-cause mortality at Day 60 and Day 90
Time Frame: Day 60 and Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
Number analyzed (Participants) | 48 | 48
Participants
  Day 60 | 8 | 5
  Day 90 | 8 | 5

7. Secondary Outcome: Number of Days Alive Outside of Hospital up to Day 28
Description: Number of days alive outside of hospital up to Day 28
Time Frame: Randomization up to Day 28
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
Number analyzed (Participants) | 48 | 48
days | 16.7 [13.97 to 19.40] | 17.1 [14.37 to 19.80]

ADVERSE EVENTS:
Time Frame: From signing of informed consent until end-of-trial visit, up to 94 days
Description: Treatment-emergent adverse events (TEAE) will be defined as any AE occurring post first administration of study drug. AEs will be coded using MedDRA dictionary.
  AE collection was assessed in the Safety population (total number of subjects dosed including placebo) only 46 participants were considered at risk for AE's in the placebo arm due to 2 participants not being treated with study IP, whereas the All-Cause Mortality was assessed in the FAS population.
Arm/Group | Abivertinib With Standard of Care | Placebo With Standard of Care
All-Cause Mortality (participants affected / at risk) | 8/48 | 5/48
Serious Adverse Events (participants affected / at risk) | 9/48 | 8/46
Other Adverse Events (participants affected / at risk) | 31/48 | 24/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abivertinib With Standard of Care (N=48) | Placebo With Standard of Care (N=46)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Brain death (General disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abivertinib With Standard of Care (N=48) | Placebo With Standard of Care (N=46)
Leukocytosis (Blood and lymphatic system disorders) | 6 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Bradycardia (Cardiac disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 3 | 3
Candida infection (Infections and infestations) | 1 | 3
Pneumonia bacterial (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 4 | 2
Alanine aminotransferase increased (Investigations) | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 4
Hypotension (Vascular disorders) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Sepsis (Infections and infestations) | 3 | 0
Hepatic enzyme increased (Investigations) | 5 | 3
Acute kidney injury (Renal and urinary disorders) | 6 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT04440007/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT04440007/SAP_001.pdf